CLINICAL TRIAL: NCT01813773
Title: Treatment With Intravitreal Aflibercept Injection For Proliferative Diabetic Retinopathy, The A.C.T Study
Acronym: ACT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ophthalmic Consultants of Long Island (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THE A.C.T. STUDY
Record Dates: First submitted 2013-02-25; First posted 2013-03-19 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - IAI every 4 weeks (Experimental): Receives 5 injections of Intravitreal Aflibercept Injection (IAI) beginning Day 1, and then at weeks 4, 8, 12, and 16. Following the 5 initial injections, this group will continue to receive IAI every 4 weeks, beginning week 20, through week 48.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI)
- Group B - IAI every 8 weeks (Experimental): Receives 5 injections of Intravitreal Aflibercept Injection (IAI) beginning Day 1, and then at weeks 4, 8, 12, and 16. Following the 5 initial injections, this group will receive IAI every 8 weeks, beginning week 24, through week 48.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI)

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection (IAI) — EYLEA (aflibercept) is a recombinant fusion protein consisting of portions of human VEGF receptors 1 and 2 extracellular domains fused to the Fc portion of human IgG1 formulated as an iso-osmotic solution for intravitreal administration. Aflibercept is a dimeric glycoprotein with a protein molecular weight of 97 kilodaltons (kDa) and contains glycosylation, constituting an additional 15% of the total molecular mass, resulting in a total molecular weight of 115 kDa. Aflibercept is produced in recombinant Chinese hamster ovary (CHO) cells.
  Other Names: Eylea

SUMMARY:
To assess the safety of intravitreal aflibercept injection in the treatment of proliferative diabetic retinopathy (PDR) by evaluating the incidence and severity of adverse events.

DETAILED DESCRIPTION:
* Single center, open label pilot study using 2.0mg intravitreal aflibercept injection. (IAI)
* 20 subjects with active PDR to be randomized into 2 groups, i.e. groups A and B.
* Subjects in both arms will be followed-up every 4 weeks until week 52.
* The primary endpoint of the study will be at week 52.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age 18 years and older
* Retinal neovascularization secondary to diabetic retinopathy
* Best corrected visual acuity in the study eye better than 20/320 using an ETDRS chart
* In the event that either eye of a potential subject meets enrollment criteria, the worse sighted eye will be enrolled into the study. Only one eye can be enrolled in the study.

Exclusion Criteria:

* Pregnant or breast-feeding women Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study and for at least 30 days after the last administration of study drug for women and at least 90 days after the last administration for men (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD];; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

  *Contraception is not required for men with documented vasectomy.

  ** Pregnancy testing and contraception are not required for women with documented hysterectomy.
* HbA1C >10 within approximately 90 days of Screening visit
* Participation in a study of an investigational drug or device within 30 days prior to potential enrollment into the study
* Prior treatment with systemic anti-VEGF agents
* Presence of any substantial ocular disease (other than diabetic retinopathy) that may compromise vision in the study eye and /or confound interpretation of the data; e.g. substantial cataracts, advanced glaucoma, optic neuritis, optic neuropathy or atrophy, marked macular atrophy, ocular vascular occlusion, history of retinal detachment, uveitis, viral or other forms of chorioretinitis, etc.
* Prior treatment with anti-VEGF therapy in the study eye within 90 days of baseline
* Prior treatment with PRP within 60 days
* Prior treatment with IAI.
* Prior treatment with triamcinolone in the study eye within 180 days of baseline.
* Prior treatment with dexamethasone in the study eye within 30 days prior to baseline.
* Intraocular surgery (including cataract surgery) in the study eye within 60 days preceding baseline
* History of vitrectomy surgery in the study eye.
* Active intraocular inflammation (grade trace or above) in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 25 mmHg despite treatment with anti-glaucoma medication)
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 180 days of study enrollment.
* History of allergy to fluorescein, topical antibiotic, povidone iodine (Betadine) or aflibercept.
* Presence of vitreous hemorrhage that completely obstructs the view of the optic nerve (amount of vitreous hemorrhage will also be gated by 20/320 criteria)
* Presence of TRD in the study eye.
* Presence of pre-retinal fibrosis (not including epiretinal membrane)
* Unwilling to discontinue sperm bank donation for any period of time after IAI treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events of intravitreal aflibercept injection in the treatment of PDR. | The primary endpoint of the study will be at week 52.

SECONDARY OUTCOMES:
Mean change in the area of fluorescein leakage in mm2 (area of neovascularization) compared to baseline. | At Weeks 24 and 52
Proportion of subjects with complete regression of neovascularization | At Weeks 24 and 52
Mean change in ETDRS BCVA from baseline | At Weeks 24 and 52
Proportion of subjects gaining > 5 letters, > 10 letters and > 15 letters from baseline | At Weeks 24 and 52
Proportion of subjects losing > 5 letters from baseline | At Weeks 24 and 52
Mean change in retinal thickness from baseline as demonstrated by Spectral Domain OCT Imaging | At Weeks 24 and 52
Proportion of subjects without vitreous hemorrhage or pre-retinal hemorrhage | At Weeks 24 and 52
Proportion of subjects with complete avoidance of panretinal laser photocoagulation (PRP)/ additional PRP | At Weeks 24 and 52
Proportion of subjects with avoidance of vitrectomy | At Weeks 24 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Glenn L Stoller, MD, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (1):
- Ophthalmic Consultants of Long Island, Lynbrook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided